CLINICAL TRIAL: NCT04653961
Title: Evaluation of a Decision Support System for People With Diabetes Who Use Multiple Daily Insulin Injections- Feasibility and Proof of Concept Studies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); DreaMed Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC096020ctil
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Subject's glucose and insulin data will be transferred to the DreaMed Advisor Pro system. Optimization of insulin treatment plan will be done using the DreaMed Advisor Pro Decision Support System-MDI algorithm. During the feasibility segment an approval of the study physician (may override the suggestions for safety reasons) will be required prior to sending the recomendations to participants. During the Proof of Concept segment, the recomendations will be sent directly to participants. Participants will be asked to follow the tretment plan for the following 2.5 weeks.
  Interventions: Device: DreaMed Advisor Pro DSS-MDI algorithm

INTERVENTIONS:
Device: DreaMed Advisor Pro DSS-MDI algorithm — The DreaMed Advisor Pro software is a proprietary algorithm, designed to provide a comprehensive analysis of individual diabetes data which consists of glucose levels and insulin delivery history. the Advisor Pro algorithm identifies glucose patterns and their possible causes, which may hamper the patient's glucose control, and recommend on adjustment to the patient-specific insulin treatment profiles as well as suggestions for personalized diabetes management tips (such as timing of meal boluses, bolus delivery compliance and personalized glucose targets).

SUMMARY:
The study comprises of two segments: a feasibility segment and a Proof of Concept segment. The study is open label, prospective study that will include up to 72 subjects in segment 1 and up to 40 subjects in segment 2. Participants are people with Type 1 or type 2 Diabetes treated with Multiple Daily Injections ( MDI) and Self Monitoring of Blood Glucose (SMBG) or intermittent Continuous Glucose Monitoring (CGM).

The study will include screening, a 2-4-week run-in period and 10-12 weeks intervention period. Subjects will be asked to record their insulin delivery during basal/bolus insulin treatment (using dedicated apps ) and their daily activities (meals, physical activity etc.) using electronic log (implemented on Dedicated Apps), for a total period of 12-16 weeks.

The goal of this study is to evaluate the safety of a decision support system for adjustment of insulin treatment plan for people with diabetes using multiple daily injections and monitoring glucose by SMBG or intermittent CGM

ELIGIBILITY:
Inclusion Criteria:

* Documented Type 1 or Type 2 Diabetes for at least 1 year prior to study enrolment
* Aged ≥ 14 years
* HbA1c of 6.5 ≤ A1c ≤ 10%
* Using basal-bolus MDI therapy:

  1. Basal insulin: Glargine, Degludec, or detemir and up to sum of 72 units of basal insulin
  2. Bolus insulin: regular insulin, rapid analogues or ultra-rapid analogues
* Subjects willing to follow study instructions:

  1. For SMBG users (only for segment 1): measure capillary blood glucose at least 4 times a day . Document blood glucose level, insulin delivery, meals and daily activities. Wear CGM.
  2. For CGM users (FGM with a reader or real-time CGM): Use CGM according to manufacture instructions, document insulin delivery, meals and daily activities.
* Subjects using CGM or SMBG that are compatible with data transmission to the study diabetes management system (i.e. for CGM, FGM with a reader).
* Fasting glucose target is < = 180 mg/dl (T2D)
* Subjects have home computer connected to the internet.
* Subjects have a smart phone compatible with study requirements.
* Subjects willing and able to sign a written informed consent form.

Exclusion Criteria:

* An episode of diabetic keto-acidosis within the month prior to study entry and/or severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrolment.
* Concomitant diseases/ treatment that influence metabolic control or any significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patients' safety
* Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus, such as:

  * Subject has unstable or rapidly progressive renal disease or is receiving dialysis
  * Subject has active proliferative retinopathy
  * Active gastroparesis
  * Subject has loss of kidney function as measured by estimated Glomerular Filtration Rate (eGFR) <45 in the previous 3 months 4. Participation in any other interventional study 5. Female subject who is pregnant or planning to become pregnant within the planned study duration
* Subject is in the "honeymoon" phase - i.e. less than 0.5 insulin units/kg per day.
* Drug or alcohol abuse.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Sensor glucose percentage of time in hypoglycemia below 54 mg/dl | 12-16 weeks
Sensor glucose percentage of time in hyperglycemia above 250 mg/dl | 12-16 weeks

SECONDARY OUTCOMES:
Percentage of readings within range of 70-180 mg/dl | 12-16 weeks
Change in HbA1C post study treatment | 12-16 weeks
Number of Serious Adverse Events | 12-16 weeks

OTHER OUTCOMES:
Percentage of readings above 180 mg/dl | 12-16 weeks
Percentage of readings below 70 mg/dl | 12-16 weeks
Mean sensor glucose | 11 weeks
Glucose variability | 12-16 weeks
Number of recommendations for changes in the treatment plan per patient | 12-16 weeks
Number of recommendations for changes in the treatment plan per iteration | 12-16 weeks
Number of physician overrides of the study system recommendations segment 1 only | 12-16 weeks
Number of physician overrides of the study system recommendations | 12-16 weeks
Total insulin dose | 12-16 weeks
The amount of basal insulin dose | 12-16 weeks
The amount of bolus insulin dose | 12-16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, MD, Study Director — Rabin Medical Center; Revital Nimri, MD, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - schneider children medical center of Israel, Petah Tikva
  - Rabin Medical Center- Belinson, Petah Tikva

IPD SHARING:
Plan to Share IPD: No